CLINICAL TRIAL: NCT01299402
Title: A Pilot Double-Blind Crossover Study on the Effects of Soulera Herbal Blend Intake on Chronic Stress and Its Biomarkers in Healthy Adults
Brief Title: A Study on the Effects of Soulera Herbal Blend Intake on Chronic Stress in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial Reasons
Sponsor: Joseph Pergolizzi, MD (Industry)
Collaborators: LeraPharm Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Pergolizzi, MD, Principal Investigator, NEMA Research, Inc.
Organization: NEMA Research, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Adaptogen Study 002
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soulera Herbal Blend (Experimental)
  Interventions: Dietary Supplement: Soulera Herbal Blend
- Placebo Blend (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soulera Herbal Blend — This a powder blend of various reputed adaptogenic herbs. The dosage will be one 8.6 gram powder sachet daily.
  Arms: Soulera Herbal Blend
Dietary Supplement: Placebo — The placebo will be a similar tasting and looking powder blend as the Soulera Herbal Blend. The dosage will be 8.6 grams per sachet daily.
  Arms: Placebo Blend

SUMMARY:
The purpose of the study was designed to evaluate the efficacy and safety of Soulera herbal mix in powder form and its effects on anxiety and the biomarkers for chronic stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 21-65.
* No concerns that would confound the study as determined by study physicians.
* Women must not be pregnant or become pregnant for the duration of the study.

Exclusion Criteria:

* The subject has a history of hypersensitivity to any of the compounds used in the study
* The subject is pregnant or breast feeding. Note: If the potential subject is a post-menarche female, a urine pregnancy test must be performed within 24 hours prior to study drug administration and confirmed negative in order for the potential subject to eb enrolled.
* History of Psychiatric Illness or Chronic Stress or Anxiety
* Hypertension, cardiovascular disease, liver, hypokalemia, or kidney disease or other health concerns that the study physician feels may confound study results
* Individuals who are cognitively impaired or who are not able to give informed consent
* Any routine prescription medication that the study physician feels may cause drug interaction with Soulera or alter the prescription medications' activity
* Previous participation in a clinical research trial within 30 days prior to randomization
* The subject has an ongoing abuse of illicit substances, alcohol, or actively smoking marijuana
* The subject uses or has used in the past 30 days any steroid formulation, be it topical like face cream, ocular as in an eye drop, nasal as in a spray, injection or pill.
* The subject is a current smoker or uses tobacco products such as chewing tobacco.
* The subject is actively engaging in the use of Herbal Medicine, Traditional Chinese Medicine, Ancient Indian Medicine, Yoga, or Ayurveda
* The subject is a night-shift worker and therefore presumably has an altered cortisol diurnal rhythm and is also unable to comply with the required cortisol collection times of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol Levels | 14 Weeks
  Change in salivary cortisol as stress biomarkers for the chronic stress response following Soulera Herbal Blend intake

SECONDARY OUTCOMES:
Change in chronic stress | 6 times during 14 weeks
  The State-Trait Anxiety Test will be given to measure the change in both chronic stress and anxiety.(
Quality of Life Questionaire | 6 times during 14 weeks
  A survery to measure your quality of life.
Spot Urine Potassium Test | 6 times during 14 weeks
  A spot urine test will be conducted to determine potassium level. Only the potassium will be measured in the urine.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Pergolizzi, Jr., M.D., Principal Investigator — NEMA Research, Inc.; Robert Taylor Jr., Ph.D., Principal Investigator — NEMA Research, Inc.; Ismail Shalaby, M.D., Ph.D., Study Director — NEMA Research, Inc.
Locations (1):
- NEMA Research, Inc., Naples, Florida, United States

REFERENCES:
- See also: Related Info — http://www.nemaresearch.com